CLINICAL TRIAL: NCT00964457
Title: Treatment of Patient With Advanced Rectum Cancer With Capecitabine and Oxaliplatin Before Under and After Radiation and With Adding Cetuximab to K_RAS Wild-type Patients.
Brief Title: Treatment of Patients With Advanced Rectum Cancer With Capecitabine and Oxaliplatin Before, Under and After Radiation and With Adding Cetuximab to K-RAS Wild-type Patients
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Copenhagen University Hospital at Herlev (Other)
Responsible Party: Ole Larsen, MD, Herlev hospital, hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GI0905
Record Dates: First submitted 2009-08-21; First posted 2009-08-25 (Estimated); Last update posted 2009-08-25 (Estimated); Status verified 2009-08

CONDITIONS: Rectum Cancer
Keywords: cetuximab; rectum cancer; radiation; MRI
MeSH Terms: conditions — Rectal Neoplasms | interventions — Cetuximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Capecitabine, oxaliplatin (Active Comparator)
  Interventions: Drug: cetuximab
- capecitabine, oxaliplatin and cetuximab (Active Comparator): capecitabine, oxaliplatin ane cetuximab
  Interventions: Drug: cetuximab

INTERVENTIONS:
Drug: cetuximab — cetuximab 500mg per meter square every second week

SUMMARY:
response rate to adding cetuximab, oxaliplatin and capecitabine to radiation for advanced rectum cancer

DETAILED DESCRIPTION:
Dynamic MRI will be used to monitor the effect of the treatment and will be compared to pathologic results.

ELIGIBILITY:
Inclusion Criteria:

* advanced rectum cancer

Exclusion Criteria:

* prior radiation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2009-08; Primary Completion 2012-07 (Estimated); Study Completion 2017-07 (Estimated)

PRIMARY OUTCOMES:
response rate | 3 years

CONTACTS AND LOCATIONS:
Locations (1):
- Herlev Hospital, Herlev, Denmark